CLINICAL TRIAL: NCT05220761
Title: FAM-CAPD: Family Assessment of Pediatric Delirium
Brief Title: Family Assessment of Pediatric Delirium
Acronym: FAM-CAPD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Laurie Lee, Adjunct Clinical Associate, University of Calgary
Other Study IDs: REB 20-2149
Record Dates: First submitted 2021-06-03; First posted 2022-02-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cornell Assessment of Pediatric Delirium — Cornell Assessment of Pediatric Delirium is a diagnostic test for PICU delirium State Behavioral Scale and Richmond Agitation and Sedation Scale are diagnostic tests for sedation and agitation in children
  Other Names: State Behavioral Scale; Richmond Agitation and Sedation Scale

SUMMARY:
In this study the investigators will assess the validity, reliability and acceptability of utilizing family members to complete a delirium screen using the Cornell Assessment of Pediatric Delirium (CAPD).

DETAILED DESCRIPTION:
Diagnosing delirium in the heterogenous PICU population is difficult. There is significant variability in pre-morbid neurodevelopmental status in children due to both age-related development as well as pre-morbid cognitive delay. The Cornell Assessment of Pediatric Delirium (CAPD) has been validated in children of all ages and developmental stages. Several confounding factors have been identified that decrease the specificity of delirium detection and include confounding syndromes (i.e. iatrogenic withdrawal syndrome), pre-existing neuro-cognitive delay, and the specialty, experience and training of the assessor. Furthermore, pediatric critical care nurses have many competing interests in prioritizing care for their patients and can struggle with trying to familiarize themselves with the concept of delirium. This is a recognized barrier to routine compliance with delirium screening in PICUs. Family screening may be extremely valuable in early identification of delirium. This has been demonstrated in the critically ill adult population, however, with respect to family detection of delirium in their own children, the reliability of a pediatric screening tool has not been evaluated.

The proposed work is designed to improve both processes of care, by improving delirium screening, and patient outcomes by engaging families in the identification, prevention and management of delirium, in critically ill children.

This study will be conducted at 2 academic PICUs in Canada. Eligible children will be consented and enrolled. Parents/caregivers will be given brief education on delirium assessment and then complete a family tool based on the Cornell Assessment of Pediatric Delirium (CAPD). This will then be validated against the RN completed CAPD.

In order to also assess the acceptability of family detection of PICU delirium interviews of family members and focus groups of HCP will be conducted using qualitative methodology to determine acceptance and feasibility and to guide future knowledge translation work.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Alberta Children's Hospital or McMaster Children's Hospital PICU during study enrollment period
* Anticipated length of stay in PICU >/=48 hours
* Substitute decision maker with the ability to provide informed consent
* Primary caregiver available for CAPD assessments,
* Primary caregiver is defined as the person primarily responsible for the care and upbringing of a child and could include: Parents, designated older sibling, foster parents/guardians, or grandparents, who fulfill this definition. There may be more than one primary caregiver for each child
* Translated CAPD and educational materials available in primary spoken language (French, Chinese, Italian or Spanish)

Exclusion Criteria:

I. Anticipated discharge/transfer within 24 hours II. Family member unable to understand the instructions for CAPD assessment

a. This will be identified by the research assistant in collaboration with the bedside care team. i.e. language/cognitive barrier III. Child in irreversible coma (i.e. persistent vegetative state, RASS -4/SBS -2 or less and not reversible)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to 2 PICUs in Canada with an expected length of stay of >/= 48 hours
Sampling Method: Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Validity of delirium screening by caregivers | 1-28 days
  Evaluate the validity of delirium screening by family or caregivers using the cornel assessment of pediatric delirium on their own children while they are admitted to a PICU

SECONDARY OUTCOMES:
Healthcare professional acceptability of family administered delirium assessment | Up to 1 year
  Explore health care professionals perception and acceptability of family administered delirium assessment in critically ill children
Family/caregiver acceptability of family administered delirium assessment | Up to 1 year
  Explore family member/caregiver perception and acceptability of family administered delirium assessment in critically ill children
Correlation between absolute score of Richmond Agitation and sedation Scale and State Behavioral Scale. | 1-28 days
  To assess the correlation between the absolute score of the Richmond Agitation and Sedation Scale [-5(unarousable) to +4(Combative)] and the State Behavioral Scale [-3 (unresponsive) to +2(agitated)] for each child in assessing sedation and agitation in critically ill children

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A. Lee, MN, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Laurie A. Lee, Calgary, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No